CLINICAL TRIAL: NCT04165278
Title: Effects of Hyperthermic Baths on Motor Symptoms of Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20190926-05
Record Dates: First submitted 2019-11-14; First posted 2019-11-15 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; temperature; hyperthermic baths; physiotherapy
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: a self-control study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hyperthermic baths (Experimental): On the first, third and fifth day of the first week, each subject will take the Hyperthermic Baths (HTB) at the same time. They will receive subjective measures before and after HTB. In the second week, no subjects accepted any intervention. On the fifteenth, seventeenth and nineteenth days of the third week, these subjects will receive two subjective measures without HTB in the same environment and scoring time as the experimental group.
  Interventions: Other: hyperthermic baths

INTERVENTIONS:
Other: hyperthermic baths — Taking hyperthermic baths

SUMMARY:
The aim of this study is to further evaluate the effects of seasonal variation and the aquatic thermal environment of hyperthermic baths (HTB) on the Motor Symptoms (MS) of Parkinson's Disease (PD), and whether the environmental temperature is associated with these effects.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all participants will give written informed consent. All participants who meet the inclusion criteria will undergo a complete history and physical examination, including an assessment using the Movement Disorder Society-United Parkinson's Disease Rating Scale (MDS-UPDRS), H&Y stage, MMSE and MOCA. Each participant will receive two subjective measures (the Movement Disorder Society-United Parkinson's Disease Rating Scale part III motor examination total scores and the modified Webster Symptoms Score) nine times in an open medication state (open state). Each participant will take hyperthermic baths (HTB) at the same time on the first, third and fifth days. The participants will receive subjective measures before and after the HTB. The time at which the subjective measures begin after the HTB will be recorded. In the second week, no participants accept any intervention. To avoid the effects of fluctuations in dopaminergic drugs concentrations, subjective measures will be given without HTB at the recorded times on the fifteenth, seventeenth and nineteenth days.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Diagnosis of Idiopathic Parkinson's Disease（IPD）based on the Movement Disorder Society clinical diagnostic criteria for Parkinson's Disease
* Subjective feeling that Motor Symptoms（MS）of Parkinson's Disease （PD） were affected by seasonal variation (i.e., MS were more severe in winter than in summer) and improved after HTB
* No change in the patient's PD medication regimen during the study

Exclusion Criteria:

* Symptomatic bradycardia, severe postural hypotension, symptomatic coronary insufficiency, severe organic heart damage, severe cerebrovascular disease, and active psychosis
* Dementia (Mini-Mental State Examination (MMSE) < 24 and Montreal Cognitive Assessment (MOCA) < 26)
* Failure to cooperate with the study requirements and poor compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-10-18 (Actual); Study Completion 2019-10-18 (Actual)

PRIMARY OUTCOMES:
The Influence of Hyperthermic Baths on Motor Symptoms as Assessed by the MDS-UPDRS Part III Motor Examination Total Scores Rating Scale | 3 week
  The minimum and maximum values of Movement Disorder Society - United Parkinson's Disease Rating Scale (MDS-UPDRS) part III motor examination total scores are 0 and 132 respectively, and higher scores mean a worse outcome.
The Influence of Hyperthermic Baths on Motor Symptoms as Assessed by the Modified Webster Symptoms Score | 3 week
  The minimum and maximum values of Modified Webster Symptoms Score are 0 and 30 respectively, and higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Yingdong Zhang, PhD, Study Director — Nanjing Medical University
Locations (1):
- Yingdong Zhang, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
we'll share our study design and the study results with other researchers
Supporting Information: Study Protocol, SAP
Time Frame: the data will become available 12 months after the study finished for 1 year
Access Criteria: clinical doctors